CLINICAL TRIAL: NCT03675217
Title: Physical Exercise Program for Family Caregivers of Dependent Patients: Randomized Clinical Trial in Primary Health Care
Brief Title: Physical Exercise Program for Family Caregivers of Dependent Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion para la Investigacion y Formacion en Ciencias de la Salud (Other)
Collaborators: Castilla-León Health Service (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GRS/VAE5-15
Record Dates: First submitted 2018-09-14; First posted 2018-09-18 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-08

CONDITIONS: Caregiver; Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Outcomes Assessor
Masking Description: Patients evaluator and Outcomes Assessor are masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PE and PCFPC (Experimental): Physical Exercise and primary care family caregivers program
  Interventions: Other: PE; Other: Usual Care
- Usual Care (Active Comparator): Usual Care: PCFPC (primary care family caregivers program)
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: PE — Physical exercise program for familiy caregivers. 36 session physical exercise (3 sessions/week) performed by physioterapist. It incluided exercices to improve coordination, aerobic capacity, control motor and strenght
  Arms: PE and PCFPC
Other: Usual Care — Usual Programe in primary care for family caregivers. 4 session (2 session/week). It incluides: ergonomy, postural hygiene, mobilitation of patients and self-care.

SUMMARY:
This estudy evaluates the effects of physical exercise program on health related quality of life (HRQoL), pain and physical fitness in family caregiver.

DETAILED DESCRIPTION:
Justification: Research indicates that the dependent patient caregiver´s have physical, psychological and social repercussions, as consequence of the care that they provide. From Primary Health Care there is a "caregiver care program" to prevent and palliate this situation, consisting mainly in education programs in care and psychotherapy. There is controversy about the effectiveness of these programs, being necessary to develop new therapeutic strategies.

Objectives: to determine the effects of a physical exercise program, adressed by the primary health care physioterapist, on health related quality of life (HRQol), pain and physical fitness in dependent patient caregivers included in the " caregiver care program" of a basic health area.

Methodology: randomized clinical trial, with control group (GC = 32) and intervention group (GI = 36), double blind and pre and post-intervention evaluation. The GC received the usual program of the " caregiver care program". The GI also carried out a multi-component exercise program for 12 weeks, with 3 weekly sessions realized in group and monitored by physiotherapists. The outcomes variables are measured by Quality of life (SF-36), Burden (Zarit), anxiety (Goldberg Ansiety Questionanaire), depression (Yesavage Questionnaire), pain intensity (EVA), disability (Roland Morris) and physical fitness (battery of fitness tests). Patients evaluator and Outcomes Assessor are masked.

Applicability of results: If the physical exercise program, carried out from the primary health care physiotherapy, improves the HRQol, pain and physical fitness, this intervention could be an effective therapeutic strategy in the "caregiver care programs". Furthermore the proposed intervention is simple, reproducible and requires few resources.

ELIGIBILITY:
Inclusion Criteria:

* Status as family caregiver and to be incluided in the "Caregiver care Program".
* Provided care to family dependent al least 6 months.
* Accept to participate in the study and sign the informed consent.
* No changes in medication for at least 3 months prior to study entry.

Exclusion Criteria:

* People whith associated pathologies that make it impossible to perform physical exercise program (moderate-intensity exercise).
* To be incluiding in other family care program
* Participation in any regular physical activity program.
* To have a formal caregiver to care for the dependent family member

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2015-09-14 (Actual); Primary Completion 2016-06-20 (Actual); Study Completion 2016-06-20 (Actual)

PRIMARY OUTCOMES:
Change in Health-related Quality of Life at different time point | Change from baseline to post-treatment (16 weeks from baseline).
  Medical Outcomes Study 36-Item Short-Form Health Survey (SF-36) V2. Spanish version. The SF-36 is a 36- item scale constructed to survey health status and quality of life. It yields an 8-scale profile of functional health and well-being scores as well as psychometrically-based physical and mental health summary. Each scale is directly transformed into a 0-100 scale. Higher scores indicate better overall quality of life.

SECONDARY OUTCOMES:
Change in burden caregiver at different time points | Change from baseline to post-treatment (16 weeks from baseline).
  Zarit Carer Burden Interview. Spanish Version. It´s a questionnaire that evaluates carer burden and asks about many commonly reported difficulties faced by carers (intraclass correlation coefficient = .71). This questionnaire presents 22 Likert-type questions each of which has a score of 0 to 4. The total score can be from 0 to 88. Higher values indicate greater burden caregiver.
Changes in anxiety at different time points | Change from baseline to post-treatment (16 weeks from baseline).
  Goldberg Anxiety Scale. Spanish version. It´s a self-reported measure that contains 9 questions designed to assed people anxiety. Scores range from 0-9. A higher score indicates a higher level anxiety
Changes in depression | Change from baseline to post-treatment (16 weeks from baseline).
  The 15-item abbreviated version of the Geriatric Depression Scale (GDS), which measures depression (internal consistency, Cronbach's α = .80). A score of 4 or more has been reported to indicate clinical signs of depression.
Change in pain assesment at different simple points | Change from baseline to post-treatment (16 weeks from baseline).
  Visual analog scale (VAS). The Vas is a 100 mm long horizontal line ranging from "0: no pain at all" on one end to "100: worst pain imaginable" on the other end. Participants mara a point along the line that best represents the pain they are experiencing at that moment. A higher score indicates a higher level of pain
Change in disability | Change from baseline to post-treatment (16 weeks from baseline).
  Roland-Morris Disability Questionnaire (RMDQ).Spanish version. It is a self-administered disability questionnaire consisting of 24 questions that are specifically related to physical functions that may be affected by back pain. Score range from 0-24. A higher score indicates a higher level of Disability
Modifications of body mass index | Change from baseline to post-treatment (16 weeks from baseline).
  Modification of the body mass index (BMI). Wheight in Kg and Height ill be combined to report BMI in kg/m^2
Changes in handgrip strength | Change from baseline to post-treatment (16 weeks from baseline).
  Handgrip strength will be assess for both hands by using a hand dynamometer (TKK 5401, Japan) and the mean value of both hands (kg*m2) is considered to be outcome.
Changes in lower extremity function | Change from baseline to post-treatment (16 weeks from baseline).
  Lower extremity function is assessed by using the "30 Second chair stand test". The patient is asked to stand upright from a standardized chair (0.43 m in height) with arms folded across the chest and to sit back down as many time as he can in 30 seconds.
Changes in postural balance | Change from baseline to post-treatment (16 weeks from baseline)
  Postural balance is assessed by performing a blind flamingo test in which the barefoot subject stood with eyes closed on one leg, while the other leg is flexed at knee leven al held at the anckle by the hand of the same side of the body. The number of trials that the subject needed to complete 30 seconds of the static position is measured. The outcomes is expressed as number of trials
Changes in flexibility | Change from baseline to post-treatment (16 weeks from baseline).
  Flexibility is assessed by using the "Sit and reach test". Here the distance between the tips of the fingers in the start to the final positions during this trunk flexion is recorded. The best result of two trials is considered the outcome.
Changes in mobility | Change from baseline to post-treatment (16 weeks from baseline).
  Mobility is assessed by using the "Timed Up and Go test". This test involves getting out of a chair, walking 3 meters to and around a cone, and returning to the chair in the shortest time possible. The best score of two trials is recorded.
Changes in maximal oxygen uptake (Vo2 max) | Change from baseline to post-treatment (16 weeks from baseline).
  Maximal oxygen uptake (Vo2 max) is assessed using the "2km Walking test " We perform the test based on the guidelines of the Afisal-Inefc Battery. For this purpose, a circuit is designed, is also used stopwatch (portable digital brand Oregon Scientific®, model SL929 Hockenheim Nero) with a precision of tenths of a second (0.1 sg) and heart rate monitors (Polar RS800 CX) to measure the heart rate at the end of the test. Procedure: The caregivers with comfortable clothes and shoes walk as fast as possible they could without running. Interpretation of the results: The time used to travel is recorded 2 kilometers, the heart rate corresponding to the end of the test expressed in beats per minute. If you spend more than 22 minutes completing the this test loses its validity. To calculate de maximal oxigen uptake (Vo2 max) this formula is used: Vo2max ( mi· kg·' ·min·' ) = 116,2 - 2,98*(time) - 0,11*(heart rate) - 0,14 (age) - 0,39*( body mass index)

CONTACTS AND LOCATIONS:
Overall Officials: Federico Montero Cuadrado, Principal Investigator — Castilla-Leon Health Service
Locations (1):
- Gerencia de Atención Primaria Valladolid-Este, Valladolid, Valladlid, Spain

IPD SHARING:
Plan to Share IPD: No